CLINICAL TRIAL: NCT04092647
Title: A Randomized Placebo-controlled Trial of Ashwagandha (Withania Somnifera) for Cognitive Dysfunction Associated With Cancer Chemotherapy.
Brief Title: Ashwagandha for Cognitive Dysfunction
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sutter Health (Other)
Responsible Party: Principal Investigator, Deepti Behl, Principal Investigator, Sutter Health
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: SIMR_onc19_IIS_Behl_Ashwaga
Record Dates: First submitted 2019-07-08; First posted 2019-09-17 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Chemo Fog
Keywords: ashwagandha; cognitive dysfunction; cancer chemotherapy
MeSH Terms: conditions — Chemotherapy-Related Cognitive Impairment; Cognitive Dysfunction | interventions — Ashwagandha

STUDY DESIGN:
Intervention Model Description: This is a 1:1 randomized double blinded placebo controlled trial.
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ashwagandha (Experimental): Ashwagandha
  Interventions: Drug: Ashwagandha
- placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ashwagandha — Ashwagandha 350 mg po BID
  Arms: ashwagandha
Drug: Placebo — Placebo 350 mg po BID
  Arms: placebo

SUMMARY:
This is a 1:1 randomized double blinded placebo controlled trial. • To determine if ashwagandha can improve cognitive dysfunction when compared with placebo in patients undergoing chemotherapy for cancer.

DETAILED DESCRIPTION:
Patients are eligible if they are currently undergoing chemotherapy or treatment with chemotherapy in the past year and state that they notice thinking or memory problems. Patients will be given FACT-Cog PCI (Version 3). Patients that score less than 63, a score that reflects moderate to severe cognitive problems, are confirmed eligible. Subjects will be randomized 1:1 in blocks of 4.

Thyroid hormone testing will be conducted at baseline and at the end of week 6 for patients with a history of thyroid disease.

Patients will receive ashwagandha 350 mg po BID or placebo. The investigators and participants will be blinded to group assignment.

Endpoint testing including the FACT-Cog PCI and total score, Hopkins verbal learning test, trail making test (abstraction and executive function), and Mini Mental Status Exam (MMSE) will be administered at baseline and after 9 weeks of treatment. Six months after stopping the study, patients will receive a link to a REDCap database to complete the FACT-Cog and state whether they used ashwagandha once they completed the study.

Active study participation will be for 9 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years and older
2. English speaking
3. Currently undergoing chemotherapy or treatment with chemotherapy in the past year
4. Self-reported memory loss, attention, visual-spatial functioning, reasoning, or information processing or cognitive changes in the first 2 cycles of chemotherapy and score < 63 on the FACT-Cog PCI
5. Able to follow instructions for testing and comply with testing
6. Able to swallow pills

Exclusion Criteria:

1. Undergoing treatment for any hormone dependent cancer
2. Planned surgical treatment
3. History of pre-existing dementia, untreated depression, psychiatric disorder, prior brain radiation or brain injury
4. History of hypotension
5. Active autoimmune disease
6. Brain metastasis
7. Taking any drugs daily that would alter cognition
8. Concurrent use of benzodiazepenes or other sedatives
9. Concurrent use of supplements that can cause sedation such as 5-HTP, calamus, California poppy, hops, Jamaican dogwood, kava, St.John's Wort, skullcap, valerian, yerba mansa
10. Currently taking hypoglycemic medications
11. History of substance abuse
12. Current or recent diagnosis of stomach ulcer or gastritis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
FACT-Cog PCI | 9 weeks
  The Functional Assessment of Cancer Therapy - Cognition (FACT-Cog) is a 37-item questionnaire designed to assess cognitive complaints in patients with cancer. The Perceived Cognitive Impairment (PCI) subscale consists of 20 items designed to measure perceived impairment in quality of life. Scores range from 0-72 where higher scores indicate less impairment and better quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Deepti Behl, MD, Principal Investigator — Sutter Health; Carol Parise, PhD, Study Director — Sutter Health
Locations (1):
- Sutter Cancer Center, Sacramento, California, United States

REFERENCES:
- [Background] Janelsins MC, Heckler CE, Peppone LJ, Kamen C, Mustian KM, Mohile SG, Magnuson A, Kleckner IR, Guido JJ, Young KL, Conlin AK, Weiselberg LR, Mitchell JW, Ambrosone CA, Ahles TA, Morrow GR. Cognitive Complaints in Survivors of Breast Cancer After Chemotherapy Compared With Age-Matched Controls: An Analysis From a Nationwide, Multicenter, Prospective Longitudinal Study. J Clin Oncol. 2017 Feb 10;35(5):506-514. doi: 10.1200/JCO.2016.68.5826. Epub 2016 Dec 28. PMID 28029304
- [Background] Ahles TA, Saykin AJ, Furstenberg CT, Cole B, Mott LA, Skalla K, Whedon MB, Bivens S, Mitchell T, Greenberg ER, Silberfarb PM. Neuropsychologic impact of standard-dose systemic chemotherapy in long-term survivors of breast cancer and lymphoma. J Clin Oncol. 2002 Jan 15;20(2):485-93. doi: 10.1200/JCO.2002.20.2.485. PMID 11786578
- [Background] Inagaki M, Yoshikawa E, Matsuoka Y, Sugawara Y, Nakano T, Akechi T, Wada N, Imoto S, Murakami K, Uchitomi Y. Smaller regional volumes of brain gray and white matter demonstrated in breast cancer survivors exposed to adjuvant chemotherapy. Cancer. 2007 Jan 1;109(1):146-56. doi: 10.1002/cncr.22368. PMID 17131349
- [Background] Wefel JS, Saleeba AK, Buzdar AU, Meyers CA. Acute and late onset cognitive dysfunction associated with chemotherapy in women with breast cancer. Cancer. 2010 Jul 15;116(14):3348-56. doi: 10.1002/cncr.25098. PMID 20564075
- [Background] Hardy SJ, Krull KR, Wefel JS, Janelsins M. Cognitive Changes in Cancer Survivors. Am Soc Clin Oncol Educ Book. 2018 May 23;38:795-806. doi: 10.1200/EDBK_201179. PMID 30231372
- [Background] Lawrence JA, Griffin L, Balcueva EP, Groteluschen DL, Samuel TA, Lesser GJ, Naughton MJ, Case LD, Shaw EG, Rapp SR. A study of donepezil in female breast cancer survivors with self-reported cognitive dysfunction 1 to 5 years following adjuvant chemotherapy. J Cancer Surviv. 2016 Feb;10(1):176-84. doi: 10.1007/s11764-015-0463-x. Epub 2015 Jul 1. PMID 26130292
- [Background] Tong T, Pei C, Chen J, Lv Q, Zhang F, Cheng Z. Efficacy of Acupuncture Therapy for Chemotherapy-Related Cognitive Impairment in Breast Cancer Patients. Med Sci Monit. 2018 May 8;24:2919-2927. doi: 10.12659/MSM.909712. PMID 29735975
- [Background] Kaur T, Kaur G. Withania somnifera as a potential candidate to ameliorate high fat diet-induced anxiety and neuroinflammation. J Neuroinflammation. 2017 Oct 12;14(1):201. doi: 10.1186/s12974-017-0975-6. PMID 29025435
- [Background] Kuboyama T, Tohda C, Komatsu K. Effects of Ashwagandha (roots of Withania somnifera) on neurodegenerative diseases. Biol Pharm Bull. 2014;37(6):892-7. doi: 10.1248/bpb.b14-00022. PMID 24882401
- [Background] Gupta M, Kaur G. Aqueous extract from the Withania somnifera leaves as a potential anti-neuroinflammatory agent: a mechanistic study. J Neuroinflammation. 2016 Aug 22;13(1):193. doi: 10.1186/s12974-016-0650-3. PMID 27550017
- [Background] Pingali U, Pilli R, Fatima N. Effect of standardized aqueous extract of Withania somnifera on tests of cognitive and psychomotor performance in healthy human participants. Pharmacognosy Res. 2014 Jan;6(1):12-8. doi: 10.4103/0974-8490.122912. PMID 24497737
- [Background] Chengappa KN, Bowie CR, Schlicht PJ, Fleet D, Brar JS, Jindal R. Randomized placebo-controlled adjunctive study of an extract of withania somnifera for cognitive dysfunction in bipolar disorder. J Clin Psychiatry. 2013 Nov;74(11):1076-83. doi: 10.4088/JCP.13m08413. PMID 24330893
- [Background] Choudhary D, Bhattacharyya S, Bose S. Efficacy and Safety of Ashwagandha (Withania somnifera (L.) Dunal) Root Extract in Improving Memory and Cognitive Functions. J Diet Suppl. 2017 Nov 2;14(6):599-612. doi: 10.1080/19390211.2017.1284970. Epub 2017 Feb 21. PMID 28471731
- [Background] Biswal BM, Sulaiman SA, Ismail HC, Zakaria H, Musa KI. Effect of Withania somnifera (Ashwagandha) on the development of chemotherapy-induced fatigue and quality of life in breast cancer patients. Integr Cancer Ther. 2013 Jul;12(4):312-22. doi: 10.1177/1534735412464551. Epub 2012 Nov 9. PMID 23142798
- [Background] Panda S, Kar A. Changes in thyroid hormone concentrations after administration of ashwagandha root extract to adult male mice. J Pharm Pharmacol. 1998 Sep;50(9):1065-8. doi: 10.1111/j.2042-7158.1998.tb06923.x. PMID 9811169
- [Background] Panda S, Kar A. Withania somnifera and Bauhinia purpurea in the regulation of circulating thyroid hormone concentrations in female mice. J Ethnopharmacol. 1999 Nov 1;67(2):233-9. doi: 10.1016/s0378-8741(99)00018-5. PMID 10619390
- [Background] Sharma AK, Basu I, Singh S. Efficacy and Safety of Ashwagandha Root Extract in Subclinical Hypothyroid Patients: A Double-Blind, Randomized Placebo-Controlled Trial. J Altern Complement Med. 2018 Mar;24(3):243-248. doi: 10.1089/acm.2017.0183. Epub 2017 Aug 22. PMID 28829155